CLINICAL TRIAL: NCT04357392
Title: Study on the Effect of Glucocorticoid Intervention on the Improvement of Blood Glucose in Patients With Exogenous Insulin Antibody Syndrome
Brief Title: Effect of Glucocorticoid on Exogenous Insulin Antibody Syndrome
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: chenfengling (Other)
Responsible Party: Sponsor-Investigator, chenfengling, Chief physician, Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University
Organization: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EIAS2020V4
Record Dates: First submitted 2020-04-19; First posted 2020-04-22 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Insulin; HbA1c; Exogenous Insulin Antibody Syndrome; Glucocorticoids
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Insulin Resistance | interventions — Prednisone; Hypoglycemic Agents; Insulin

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, single center, pragmatic clinical trial
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glucocorticoid intervention group (Experimental): prednisone
  Interventions: Drug: Prednisone
- Placebo control group (Placebo Comparator): placebo
  Interventions: Drug: Prednisone

INTERVENTIONS:
Drug: Prednisone — Prednisone 10mg, TID * 2 weeks, decreasing 5mg per week, continuous treatment for 8 weeks
  Other Names: oral antidiabetic agents; insulin

SUMMARY:
Diabetic patients who have long-term insulin used can product antibody against exogenous insulin, the investigators named this condition Exogenous insulin antibody syndrome (EIAs). Exogenous insulin antibody can cause blood glucose fluctuation, high blood glucose and refractory hypoglycemia, and have a serious impact on the health of diabetic patients. After adding glucocorticoid, some EIAs patients can reduce insulin dosage, correct hypoglycemia, even eliminate insulin antibody in about half a year, and achieve the goal of blood glucose stability. But up to now, there is no study to evaluate the improvement of blood glucose by glucocorticoid intervention in EIAS patients receiving insulin therapy. This project plans to collect 20 cases of EIAS and carry out a randomized, double-blind, placebo-controlled clinical trial to evaluate the improvement of blood glucose by glucocorticoid intervention.

DETAILED DESCRIPTION:
Diabetic patients who have long-term insulin used can product antibody against exogenous insulin, the investigators named this condition Exogenous insulin antibody syndrome (EIAs).Exogenous insulin antibody can lead to serious clinical consequences , such as blood glucose fluctuations, high blood glucose and refractory hypoglycemia, which is not only affect patients' blood glucose control, but also have a serious impact on the health of diabetic patients. Change to the oral antidiabetic drugs, change the insulin type or add glucocorticoids to the patients with serious disease are the main treatments. However, most of these treatment schemes are case reports, and there is no randomized controlled cohort study on the treatment scheme. The biosynthetic human insulin sequence is exactly the same as that of human insulin. Why do some diabetics have insulin antibody? The investigators speculated that insulin antibody production in some patients with EIAs is related to autoimmune disorder. After adding glucocorticoid, some EIAs patients can reduce insulin dosage, correct hypoglycemia, even eliminate insulin antibody in about half a year, and achieve the goal of blood glucose stability. However, there is no study to evaluate the effect of glucocorticoid intervention on the improvement of blood glucose in the EIAs population. This project plans to collect 20 cases of EIAs and carry out a randomized, double-blind, placebo-controlled clinical trial to evaluate the improvement of blood glucose by glucocorticoid intervention, so as to provide scientific basis for the standardized diagnosis and treatment of EIAs.

ELIGIBILITY:
Inclusion Criteria:

1. The diagnosis of type 2 diabetes was in accordance with the WHO diagnostic criteria of diabetes in 1999:fasting blood glucose ≥ 7.0mmol/l and / or blood glucose ≥ 11.1mmol/l in 2 hours after OGTT
2. Aged between 30-60 years
3. Positive detection of insulin antibody, hyperinsulinemia (refer to WHO standard in 1999, fasting insulin > 15 μ IU / ml or 2h postprandial insulin > 80 μ IU / ml)
4. Type 2 diabetes mellitus patients who receiving insulin therapy
5. Those meeting all the above standards can be included

Exclusion Criteria:

1. Patients who had used animal insulin before the study
2. Type 1 diabetes, gestational diabetes and special type diabetes
3. Diabetic acute complications (ketoacidosis, hyperosmotic nonketotic coma, lactic acidosis) or serious chronic complications ; serious chronic complications (proliferative retinopathy, foot ulcer or gangrene, Complications of heart, brain and kidney)
4. Patients with other serious heart disease, endocrine disease, autoimmune or chronic wasting disease
5. Patients with severe primary diseases such as liver, kidney and hematopoietic system , Patients with psychosis
6. Patients who are using or need to use thiol containing drugs in the near future
7. Patients with severe insulin allergy
8. Glucocorticoid contraindications (severe psychosis and epilepsy, active peptic ulcer or tuberculosis, recent gastrointestinal anastomosis, fracture, wound repair period, corneal ulcer, adrenocortical hyperfunction, severe hypertension, pregnant women, infection beyond the control of antibiotics, such as varicella, mould infection, etc.)

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-05-20 (Estimated); Primary Completion 2022-05-20 (Estimated); Study Completion 2023-05-20 (Estimated)

PRIMARY OUTCOMES:
Number of patients with HbA1c <7% at 12 and 24 weeks | 24 weeks

SECONDARY OUTCOMES:
Blood glucose fluctuation at 4, 12 and 24 weeks | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chen, Principal Investigator — The Ninth People's Hospital Affiliated to Shanghai Jiaotong University

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: when summary data are published